CLINICAL TRIAL: NCT02177253
Title: A Comparison of Ipratropium Bromide/Salbutamol (40 mcg / 200 mcg, One Inhalation) Delivered by the Respimat ® Inhaler to COMBIVENT Inhalation Aerosol (Two Inhalations), Ipratropium Bromide Respimat ® and Placebo of Each Formulation in a 12-week, Double-blind, Safety and Efficacy Study in Adults With Chronic Obstructive Pulmonary Disease
Brief Title: Ipratropium Bromide/Salbutamol Delivered by the Respimat® Inhaler Compared to Ipratropium Bromide Respimat®, COMBIVENT® Inhalation Aerosol and Placebo in Adults With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.46
Record Dates: First submitted 2014-06-20; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol

ARMS (5):
- Ipratropium bromide / Salbutamol Inhalation solution (Experimental)
  Interventions: Drug: Ipratropium bromide / Salbutamol
- Placebo Inhalation solution (Placebo Comparator)
  Interventions: Drug: Placebo Inhalation solution
- Ipratropium bromide Inhalation solution (Experimental)
  Interventions: Drug: Ipratropium bromide
- COMBIVENT Inhalation Aerosol (ipratropium bromide/salbutamol) (Active Comparator)
  Interventions: Drug: COMBIVENT Inhalation Aerosol
- Placebo Inhalation Aerosol (Placebo Comparator)
  Interventions: Drug: Placebo Inhalation Aerosol

INTERVENTIONS:
Drug: Ipratropium bromide / Salbutamol
  Arms: Ipratropium bromide / Salbutamol Inhalation solution
Drug: Placebo Inhalation solution
  Arms: Placebo Inhalation solution
Drug: Ipratropium bromide
  Arms: Ipratropium bromide Inhalation solution
Drug: COMBIVENT Inhalation Aerosol
  Arms: COMBIVENT Inhalation Aerosol (ipratropium bromide/salbutamol)
Drug: Placebo Inhalation Aerosol
  Arms: Placebo Inhalation Aerosol

SUMMARY:
The primary objective of this study was to compare the long-term (12-week) bronchodilator efficacy and safety of ipratropium bromide / salbutamol combination administered by the Respimat® 40 mcg / 200 mcg (one inhalation q.i.d.) to COMBIVENT Inhalation Aerosol (two inhalations q.i.d.), ipratropium bromide Respimat® (one inhalation q.i.d.) and Placebo formulations of each in patients with Chronic Obstructive Pulmonary Disease (COPD). An additional objective was to show the superiority of Combivent Respimat as compared to ipratropium bromide (40 mcg) Respimat. Steady state pharmacokinetics over one dosing interval following four weeks of therapy were also characterized.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of COPD and the following spirometric criteria:

  * Visit 1 (Screening) and Visit 2: Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 ≤65% of predicted normal and FEV1 ≤70% of FVC
* Male or female patients 40 years of age or older
* Patients must have a smoking history of more than ten pack-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
* Patients must be able to perform pulmonary function tests and maintain records during the study period as required in the protocol
* Patients must be able to be trained in the proper use of an MDI (metered dose inhaler) and the Respimat® inhaler
* All patients must sign an Informed Consent Form prior to participation in the trial

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinically relevant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion, the patient is excluded
* All patients with a SGOT (serum glutamic oxaloacetic transaminase) >80 IU/L, SGPT (serum glutamic pyruvic transaminase) >80 IU/L, bilirubin >2.0 mg/dL or creatinine >2.0 mg/dL will be excluded regardless of the clinical condition
* Patients who have a total blood eosinophil count ≥600/mm3
* Patients with a recent history (i.e., one year or less) of myocardial infarction
* Patients with a recent history (i.e., three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy
* Patients with a history of cancer, other than treated basal cell carcinoma, within the last 5 years
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of a thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1
* Patients with a history of asthma or allergic rhinitis
* Patients with a history of and/or active alcohol or drug abuse
* Patients with known active tuberculosis
* Patients with an upper or lower respiratory tract infection or COPD exacerbation in the 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients with current significant psychiatric disorders
* Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy
* Patients who are being treated with cromolyn sodium or nedocromil sodium
* Patients who are being treated with antihistamines for any excluded allergic conditions
* Patients using oral corticosteroid medication at unstable doses (i.e., less than 6 weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Patients who initiated use of an inhaled steroid or changed doses less than 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period
* Patients who are being treated with beta-blocker medications, MAO (monoamine oxidase) inhibitors or tricyclic antidepressants. Beta blocker eye medications (e.g., Betoptic) for treatment of non-narrow angle glaucoma are allowed
* Patients who have had changes in their therapeutic plan within the last 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception
* Patients with known hypersensitivity to anticholinergic drugs or any component of the ipratropium bromide/salbutamol Respimat® solution (including BAC (Benzalkonium chloride) and EDTA (Ethylenediaminetetraacetic acid)) or the ipratropium bromide/salbutamol MDI components
* Previous participation in this study
* Patients who are currently participating in another study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1118 (Actual)
Dates: Start 2002-10; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
FEV1 TAUC0-6 (Total area under the FEV1 (forced expiratory volume in one second) curve from 0 to 6 hours divided by six) | Day 85

SECONDARY OUTCOMES:
FEV1 TAUC0-6 | Days 1, 29 and 57
FEV1 TAUC0-8 | Days 1, 29, 57 and 85
Peak FEV1 post treatment over two hours | Days 1, 29, 57 and 85
Change from baseline in Peak FEV1 response | Days 1, 29, 57 and 85
Area under the FEV1 curve from 0 to 6 hours above test-day baseline divided by six for normalization (AUC0-6) | Days 1, 29, 57 and 85
Onset of therapeutic FEV1 response | Days 1, 29, 57 and 85
Duration of therapeutic FEV1 response | Days 1, 29, 57 and 85
Time to peak FEV1 response | Days 1, 29, 57 and 85
TAUC0-6, TAUC0-8 and peak FVC (Forced vital capacity) | Days 1, 29, 57 and 85
Amount of beta agonist therapy used as rescue medication during the treatment period | up to day 85
Number of patients using concomitant medication including corticosteroids during the treatment period | up to day 85
Weekly means of daily symptom scores over the treatment period | up to day 85
Number of patients with at least one COPD exacerbation | up to day 85
Number of COPD exacerbations during the treatment period | up to day 85
Physician's Global Evaluation | Days 1, 29, 57 and 85
Trough PEFR (peak expiratory flow rate) measured by the patient at home once daily | up to day 85
Number of patients with adverse events | up to day 85
Incidence of paradoxical bronchoconstriction on the test day | up to day 85
Number of COPD exacerbation days | up to day 85
Number of patients with clinically significant changes in vital signs | Baseline, days 1, 29, 57 and 85
Number of patients with abnormal changes in laboratory parameters | Days 29 and 85
Number of patients with abnormal changes in 12-lead electrocardiogram (ECG) parameters | pre-treatment and 1 hour post-treatment on days 1, 29 and 85
Plasma ipratropium and salbutamol concentrations | pre-treatment, 5, 15, 30 and 60 minutes and 2, 4 and 8 hours after inhalation of test drug on day 29
Renal excretion amounts of ipratropium and salbutamol | 0-2 hours, 2-8 hours at day 29
Length of COPD exacerbations during the treatment period | up to day 85